CLINICAL TRIAL: NCT02914392
Title: Multi-center Clinical Study on the Relationship Between Maternal Exposure to Important Environmental Factors and Fetal Congenital Heart Disease
Brief Title: Study on the Relationship Between Maternal Exposure to Environmental Factors and Fetal Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kun Sun, Director of Department of Pediatric Cardiology, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-023
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Congenital Heart Disease
Keywords: case control study; Environmental Factors; Fetal Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The content of folic acid in serum of cases and controls is determined.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fetal congenital heart disease cases: Gravidas with fetal congenital heart disease diagnosed by fetal echocardiography
- Matched Controls for fetal congenital heart disease cases: Gravidas without fetal congenital heart disease

SUMMARY:
The objective of this study is to research the relationship between maternal exposure to environmental factors and fetal congenital heart disease in a community-based case-control study.

DETAILED DESCRIPTION:
This is a community-based case-control study in SHANGHAI,a municipality in CHINA. Cases will be identified from maternity centers. Matched controls will be accrued from the same region as the case came from. Pregnant cases and their controls are women (18-45 years). Cases are gravidas with fetal congenital heart disease diagnosed by echocardiography in 16th-29nd of gestational weeks. Controls are pregnant women without fetal congenital heart disease diagnosis. Only gravidas who are willing to have complete pregnancy checks and finally delivery or abortion in the hospital are interviewed are eligible for the study. About 2 controls matched by year of birth and region will be allocated to each case. A standardized questionnaire will be used for all cases and controls. Field investigations are also conducted for them by quantitative measurement of some chemical, physical and nutritional factors related indicators may affect fetal cardiovascular development. Study participants will be asked for their informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Gravida with singleton pregnancy taking fetal echocardiography in 16th-29nd of gestational weeks.
2. Complete pregnancy check in the hospital, and finally delivery or abortion in the hospital.
3. On the basis of informed consent，willing to cooperate with our group.

Exclusion Criteria:

1. Pregnant women with serious pregnancy complications .
2. Pregnant women suffering from mental illness, can't take care of themselves. 3) Fetus diagnosed with chromosomal abnormalities in pregnant women .

4）Repeated explanation does not cooperate in pregnant women.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Gravidas with singleton pregnancy living in SHANGHAI
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fetal Congenital heart disease | Sep 2016 to Jul 2018

CONTACTS AND LOCATIONS:
Overall Officials: Kun Sun, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - School of environmental science and engineering, Shanghai jiaotong university, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided